CLINICAL TRIAL: NCT04710121
Title: The Effect of Virtual Reality Glasses Used During Colonoscopy on Vital Signs, Pain and Anxiety Level
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Esra KILINÇ AKMAN (Other)
Responsible Party: Sponsor-Investigator, Esra KILINÇ AKMAN, Master of Science (MSC) Nurse, Istanbul University - Cerrahpasa
Organization: Istanbul University - Cerrahpasa (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2020/42-12
Record Dates: First submitted 2021-01-03; First posted 2021-01-14 (Actual); Last update posted 2021-01-14 (Actual); Status verified 2021-01

CONDITIONS: Colonoscopy
Keywords: colonoscopy; virtual reality glasses; pain; anxiety; vital signs; nursing
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: A randomized controlled study to determine the effects of virtual reality glasses used during the colonoscopy on vital signs, pain, and anxiety levels.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Experimental): The experimental group will be asked about their anxiety states with the "State and Trait Anxiety Inventory", their pain conditions with the Analog Scale (VAS), and their first life findings will be measured, and the first measurement values will be recorded in the "Vital Signs Follow-up Form". Virtual reality glasses will be placed on the patient's head during colonoscopy. The duration of the colonoscopy will vary between 3-10 minutes, videos with music background, park, nature and seaside walks, underwater videos, which the patient chooses, will be watched and the "Vital Signs Tracking Form" Second measurement values will be recorded by making measurements. Immediately after the colonoscopy procedure is completed, "Visual Analogue Scale (VAS)", "Vital Signs Follow-up Form" (measurement will be made and 3rd measurement values will be recorded. The "State Anxiety Inventory" will be read and the answers will be recorded.
  Interventions: Other: Virtual Reality Glasses
- Control Arm (No Intervention): No application will be made in the control group. during and after colonoscopy and routine treatment and care will be applied.

INTERVENTIONS:
Other: Virtual Reality Glasses — Virtual Reality Glasses (VRG), one of the methods of distracting attention; widely used in clinical medical care to relieve symptoms by providing the opportunity to create therapeutic environments for the evaluation and treatment of medical conditions. Virtual reality is a computer simulation technique that enables individuals to hear and feel the sounds and corresponding stimuli accompanying the visual image through headphones. The most basic feature that distinguishes virtual reality (VR) glasses from similar applications is that it gives individuals a real feeling. VR has helped to distract patients from mental processing and reduce the amount of pain. Virtual reality glasses, which are inexpensive to apply and use, do not cause side effects, and can be used in the recovery of the individual, are an intervention that can be preferred in nursing practices.
  Other Names: Assigned Interventions
  Arms: Intervention Arm

SUMMARY:
The study was planned as a randomized controlled experimental study to determine the effect of virtual reality glasses used during a colonoscopy on vital signs, pain, and anxiety level. After the approval of the ethics committee and institutional permission, 60 patients who applied to the endoscopy unit for colonoscopy procedure between 1 October 2020 and 1 October 2021 and met the inclusion criteria will be included in the study. Within the scope of the planned study, the sample size in the light of the reported academic studies was determined as effect size d = 0,665 (effect size), α = 0.05 (margin of error), 1-β = 0.80 (Power) and by using the G-Power package program with the specified criteria. It was decided to recruit 58 people (29 people per group). The block randomization method will be used to determine the experimental and control groups. In order for the groups to be distributed homogeneously, the order produced by a computer program (https://www.randomizer.org/) will be used. Randomization will be done by a biostatistician outside the researcher. Patients who meet the inclusion criteria and agree to participate in the study will be assigned to the experimental and control groups according to the randomization list. Before the colonoscopy, the patient will be visited and information will be given about the purpose, content, and intervention to be applied. After obtaining verbal and written consent from the patients who accepted to participate in the study, the "Individual Characteristics Form" will be filled. Then, before the colonoscopy procedure, the anxiety states of the patients in the experimental and control groups will be asked with the "State and Trait Anxiety Inventory", their pain status with the Analog Scale (VAS), and their first life findings will be measured and the first measurement values will be recorded in the "Vital Signs Follow-up Form".

The patients in the experimental group will be informed about the virtual glasses before the colonoscopy procedure and the virtual reality glasses will be placed on the patient's head during the procedure. Then, during the colonoscopy procedure, the duration of the colonoscopy will vary between 3-10 minutes, and during the colonoscopy period, videos with music background, parks, nature and seaside walks, underwater, etc., will be watched by the patient and the "Vital Signs Tracking Form" The second measurement values will be saved by making measurement to.

Immediately after the colonoscopy procedure is finished, "Visual Analogue Scale (VAS)", "Life Findings Follow-up Form" (measurement will be made and 3rd measurement values will be recorded. The "State Anxiety Inventory" will be read and the answers will be recorded. The standard application will be applied to the patients in the control group during the colonoscopy procedure and the second measurement values will be recorded by measuring the "Vital Signs Follow-up Form".Immediately after the colonoscopy procedure is completed, the third measurement value will be recorded by measuring the "Visual Analogue Scale (VAS)" and "Vital Signs Follow-up Form". "State Anxiety Inventory" will be read and the answers recorded.

DETAILED DESCRIPTION:
The universe of the research; patients who are between October 1, 2020, and October 1, 2021, in the endoscopy unit for colonoscopy procedure where the study will be conducted will comprise the patients who meet the inclusion criteria and agree to participate in the study. The research was planned as a randomized controlled experimental study. The block randomization method will be used to determine the experimental and control groups. In order for the groups to be distributed homogeneously, the order produced by a computer program (https://www.randomizer.org/) will be used. Randomization will be done by a biostatistician outside the researcher. Patients who meet the inclusion criteria and agree to participate in the study will be assigned to the experimental and control groups according to the randomization list. Research data will be collected in a hospital's endoscopy unit between 1 October 2020 - 1 October 2021. The independent variable of the study is virtual reality glasses. The dependent variables of the study are anxiety states, pain intensity, and vital signs score average. In the research, "Individual Characteristics Form", "State and Trait Anxiety Inventory", the Analog Scale (VAS), and "Vital Signs Follow-up Form" prepared by the researcher in line with the literature will be used as data collection tools.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and over,
* Having the ability to read and write in Turkish,
* According to the American Anesthesiologists Association (ASA) classification; ASA score of I or II,
* The patient expresses that he / she has no mental disorder,
* Stating that the patient is not using any anti-anxiety (anxiolytic) medication,
* Migraine, vertigo, active nausea, vomiting, headache… etc. absence of a situation,
* No vision, hearing or perception problems,
* No previous abdominal surgery (no large intestine surgery, lower abdominal surgery),
* Being conscious, oriented, cooperative and open to communication.

Exclusion Criteria:

* Malignancy (GIS and all malignancies),
* Not enough bowel cleansing,
* There is no fasting period of at least 8 hours,
* Possible pregnancy or pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2021-01-03 (Estimated); Primary Completion 2021-06-20 (Estimated); Study Completion 2021-12-20 (Estimated)

PRIMARY OUTCOMES:
Pre-colonoscopy state of anxiety | Reported state of anxiety in the first 10 minutes before the colonoscopy procedure
  The statements in the state anxiety scale were answered as "none", "a little", "a lot" and "completely" according to the person's feelings, while the statements in the continuity anxiety scale were "almost never", "sometimes", "much time" according to the frequency of emotions experienced by the person. "And" almost always ". It is 50 for State Anxiety Scale and 35 for Trait Anxiety Scale. It is scored between 20-80 in two scales. The higher the score, the higher the anxiety level. If the score obtained from the scale is 20-39, it indicates mild, 40-59 indicates moderate and 60-80 indicates severe anxiety.
Pre-colonoscopy pain severity | Reported pain severity in the first 5 minutes before the colonoscopy procedure
  Pain severity assessment with Visual Assessment Scale (VAS) Score: 0-10; 0- No Pain, 10- Worst pain
Heart rate before the colonoscopy procedure | Immediately before the colonoscopy procedure
  60 to 100 beats per minute is normal.
Blood pressure before the colonoscopy procedure | Immediately before the colonoscopy procedure
  90/60 mm Hg to 120/80 mm Hg is normal.
Respiration rate before the colonoscopy procedure | Immediately before the colonoscopy procedure
  12 to 18 breaths per minute is normal.
Oxygen saturation (SpO2) before the colonoscopy procedure | Immediately before the colonoscopy procedure
  Normal oxygen saturation usually ranges from 95 to 100%.
Heart rate during the colonoscopy procedure | During the colonoscopy procedure
  60 to 100 beats per minute is normal.
Blood pressure during the colonoscopy procedure | During the colonoscopy procedure
  90/60 mm Hg to 120/80 mm Hg is normal.
Respiration rate during the colonoscopy procedure | During the colonoscopy procedure
  12 to 18 breaths per minute is normal.
Oxygen saturation (SpO2) during the colonoscopy procedure | During the colonoscopy procedure
  Normal oxygen saturation usually ranges from 95 to 100%.
Heart rate after the colonoscopy procedure | Reported heart rate/per minute in the first 5 minutes after the colonoscopy procedure
  60 to 100 beats per minute is normal.
Respiration rate after the colonoscopy procedure | Reported respiration rate/per minute in the first 5 minutes after the colonoscopy procedure
  12 to 18 breaths per minute is normal.
Blood pressure after the colonoscopy procedure | Reported blood pressure in the first 5 minutes after the colonoscopy procedure
  90/60 mm Hg to 120/80 mm Hg is normal.
Oxygen saturation (SpO2) after the colonoscopy procedure | in the first 5 minutes after the colonoscopy procedure
  Normal oxygen saturation usually ranges from 95 to 100%.
Post-colonoscopy pain | Reported pain severity in the first 5 minutes after the colonoscopy procedure
  Pain severity assessment with Visual Assessment Scale (VAS) Score: 0-10; 0- No Pain, 10- Worst pain
Pre-colonoscopy state of anxiety | Reported state of anxiety in the first 10 minutes after the colonoscopy procedure
  The statements in the state anxiety scale were answered as "none", "a little", "a lot" and "completely" according to the person's feelings, while the statements in the continuity anxiety scale were "almost never", "sometimes", "much time" according to the frequency of emotions experienced by the person. "And" almost always ". It is 50 for State Anxiety Scale and 35 for Trait Anxiety Scale. It is scored between 20-80 in two scales. The higher the score, the higher the anxiety level. If the score obtained from the scale is 20-39, it indicates mild, 40-59 indicates moderate and 60-80 indicates severe anxiety.

SECONDARY OUTCOMES:
Satisfaction status with virtual reality glasses application | Satisfaction is reported within the first 15 minutes after the colonoscopy procedure.
  Visual Evaluation Scale (VAS) score similar satisfaction rating: 0-10; 0- nothing, 10- very good

CONTACTS AND LOCATIONS:
Overall Officials: Ayfer ÖZBAŞ, Prof, Study Director — Istanbul University - Cerrahpasa; Esra KILINÇ AKMAN, MSC, Study Chair — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul Provincial Health Directorate Prof. Dr. Cemil Taşcioğlu City Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No